CLINICAL TRIAL: NCT00000955
Title: Two-Stage Tuberculin (PPD) Skin Testing in Individuals With Human Immunodeficiency Virus (HIV) Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Warner Lambert - Parke Davis (Industry)
Responsible Party: Rona Siskind, DAIDS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CPCRA 008; 11560 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Tuberculosis; Immunologic Tests; Tuberculin; Tuberculin Test; AIDS-Related Opportunistic Infections; Injections, Intradermal; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Hypersensitivity, Delayed
MeSH Terms: conditions — HIV Infections; Tuberculosis; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Hypersensitivity, Delayed | interventions — Tuberculin

ARMS (1):
- A (Other): All eligible study participants
  Interventions: Drug: Tuberculin Purified Protein Derivative

INTERVENTIONS:
Drug: Tuberculin Purified Protein Derivative — Administered intradermally at 5 TU per 0.1 mL

SUMMARY:
To quantitate in an HIV-infected population the percentage of patients demonstrating the "booster" phenomenon (attainment of a positive response to a second tuberculin purified protein derivative skin test when the first skin test was negative); to determine the relationship between the booster phenomenon and CD4-positive lymphocyte cell counts; to detect any relationship between the booster phenomenon and HIV exposure category.

The accuracy of skin testing to detect Mycobacterium tuberculosis (MTb) infection is dependent upon the host's ability to mount a delayed-type hypersensitivity (DTH) reaction; however, the DTH response may be impaired or absent in patients with impaired cell-mediated immunity, a classic characteristic of HIV infection. Patients in whom immunity is diminished, but not absent, may test negative the first time a purified protein derivative skin test for MTb is administered, but if the same skin test is repeated, a positive DTH response may then be elicited. This occurrence is known as the "booster" phenomenon.

DETAILED DESCRIPTION:
The accuracy of skin testing to detect Mycobacterium tuberculosis (MTb) infection is dependent upon the host's ability to mount a delayed-type hypersensitivity (DTH) reaction; however, the DTH response may be impaired or absent in patients with impaired cell-mediated immunity, a classic characteristic of HIV infection. Patients in whom immunity is diminished, but not absent, may test negative the first time a purified protein derivative skin test for MTb is administered, but if the same skin test is repeated, a positive DTH response may then be elicited. This occurrence is known as the "booster" phenomenon.

Patients who have had a negative purified protein derivative (PPD) skin test for M. tuberculosis within 7-28 days prior to study entry will receive a second PPD test by the Mantoux method (5 TU intradermally to the volar aspect of the forearm). Skin tests will be read 48-72 hours after application. Patients with a positive skin test (defined as an induration, or small hard knot, of 5 mm or greater forming beneath the skin) will be referred to their primary physicians for further evaluation.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* Negative PPD skin test within previous 7-28 days.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Steroids.
* Live viral vaccines.
* Antihistamines.
* Chemoprophylaxis or chemotherapy for suspected or confirmed tuberculosis.

Patients with the following prior conditions are excluded:

* History of documented positive PPD skin test.
* History of tuberculosis or who are presently receiving chemoprophylaxis or chemotherapy for suspected or confirmed tuberculosis.
* History of sensitivity to tuberculin or components of PPD.

Prior Medication:

Excluded:

* Live viral vaccine within the past 4 weeks.
* Steroid therapy within the past 4 weeks.
* Antihistamines within the past week.
* Chemoprophylaxis or chemotherapy for suspected or confirmed tuberculosis.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Primary Completion 1992-12 (Actual); Study Completion 1992-12 (Actual)

PRIMARY OUTCOMES:
To estimate the percentage of HIV-infected individuals who demonstrate the booster effect | Throughout study

SECONDARY OUTCOMES:
To determine the relationships among the booster effect, CD4+ cell count, and other HIV-related patient characteristics | Throughout study
To determine the relationship of boosting to CD4+ cell counts, HIV exposure categories, demographics, and TB risk categories | Throughout study
To determine the relationship of induration size after the first PPD skin test to that after the second PPD skin test | After the second PPD skin test

CONTACTS AND LOCATIONS:
Overall Officials: Thompson C, Study Chair; Gordin F, Study Chair
Locations (14):
- United States (14):
  - Hill Health Corp, New Haven, Connecticut
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Clinical Directors Network of Region II, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Thompson C, Gordin F, Muth K, Daniels K, Matts J, Maiatico G, Deyton L. Two stage tuberculin (PPD) skin testing in individuals with HIV infection. Int Conf AIDS. 1992 Jul 19-24;8(3):140 (abstract no PuB 7546)
- [Background] Webster CT, Gordin FM, Matts JP, Korvick JA, Miller C, Muth K, Brown LS, Besch CL, Kumi JO, Salveson C, et al. Two-stage tuberculin skin testing in individuals with human immunodeficiency virus infection. Community Programs for Clinical Research on AIDS. Am J Respir Crit Care Med. 1995 Mar;151(3 Pt 1):805-8. doi: 10.1164/ajrccm.151.3.7881675.